CLINICAL TRIAL: NCT01361633
Title: The Cognitive Enhancing Effects of D-Cycloserine Among Non-Demented Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 126177; DIEF002352HI (Other Grant/Funding Number: Hartford Hospital)
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2019-10

CONDITIONS: Treatment; Placebo
Keywords: d-cycloserine; geriatric; neuropsychology; cognition; cognitive-enhancer; aging; neuropsychological functioning
MeSH Terms: interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication (Experimental): 250 mg d-cycloserine
  Interventions: Drug: d-cycloserine
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: d-cycloserine — single oral administration of 250 mg d-cycloserine
  Other Names: Seromycin
  Arms: Medication
Drug: Sugar Pill — Single oral administration 250 mg Sugar Pill
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
The goal of this study is to determine whether a study medication (d-cycloserine) improves the ability of older adults to perform on tests of neuropsychological functioning. Tests of neuropsychological functioning assess attention, memory, and executive functioning skills (for example, problem-solving, planning and organizing skills). It was hypothesized that participants who received study medication would perform better on neuropsychological tests than would participants who received the sugar pill.

DETAILED DESCRIPTION:
Accumulating data support the augmenting effects of d-cycloserine (DCS) when combined with exposure-based treatment for anxiety disorders. Additional research is needed to determine whether DCS facilitates other forms of cognitive processing (e.g., attention, memory, executive functioning) that are involved in cognitive behavioral therapies which do not rely on extinction as a mechanism of action. This question is particularly important among older adults who have experienced normal age-related declines in cognitive functioning, which may interfere with their ability to benefit from cognitive-behavioral therapies. The aim of the current study was to determine the cognitive enhancing effects of DCS on neuropsychological test performance among healthy older adults. It was hypothesized that participants who received d-cycloserine would demonstrate superior performance on neuropsychological tests than would participants who received placebo.

ELIGIBILITY:
Inclusion Criteria:

* age 60 or older
* native English speaker

Exclusion Criteria:

* diagnosis of current psychiatric disorder
* substance abuse past 3 months
* cognitive impairment
* neurological disorder
* poor health or unstable medical condition
* positive toxicology screen
* current use of isoniazid
* current use of trecator
* severe renal insufficiency

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen J. Diefenbach, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Anxiety Disorders Center, Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria:
  * age 60+
  * fluent in English
  Exclusion criteria:
  * current psychiatric disorder other than GAD
  * substance abuse w/in past 3 months
  * MMSE score of <24
  * neurological disorder
  * poor health or unstable medical condition
  * positive tox screen tests
  * current use of Isoniazid or Trecator
  * renal insufficiency
Pre-assignment Details: Participants were excluded at Baseline if they had abnormal lab results (6), were taking Aricept (1), were too worried about taking medication (1), or had concurrent depression (1).
Groups:
- Sugar Pill: Placebo Control
Period: Overall Study
Arm/Group | Medication | Sugar Pill
Started | 25 | 26
Completed | 19 | 23
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication | Sugar Pill | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6.73) | 70 (8.44) | 69 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: California Verbal Learning Test-II (CLVT-II)
Description: The CLVT-II is an assessment of verbal learning and memory which measures recall and recognition scores, encoding strategies, learning rates and error types. A list learning task with 16 words from 4 semantic categories are read over a series of 5 list presentations. Recall is assessed after learning and at a 20-minute delay. Software produces a report that computes raw and standardized scores. Our dependent variable was the age adjusted t-score for total number of words recalled after 5 trials. A higher score indicated better recall. The maximum possible score was 80 and a minimum was 0.
Time Frame: Outcome measures will be collected during a single neuropsychological testing administration lasting approximately 3 hours without patient follow up. Scores for the experimental and control group were compared.
Measure: Mean (Standard Deviation); unit: age adjusted t-scores
Groups:
- Medication: 250mg d-cycloserine
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 19 | 23
age adjusted t-scores | 55.84 (10.37) | 55.39 (10.73)

2. Secondary Outcome: Continuous Performance Test
Description: Sustained attention was assessed using the Penn version of the Continuous Performance Test. During the CPT the participant responds to a target stimulus (e.g., the letter "A"), while inhibiting responding to distractor stimuli. Reaction time to correct targets (true positives) was used as the dependent variable. Faster reaction times indicate better performance.
Time Frame: Outcome measures will be collected during a single neuropsychological testing administration lasting approximately 3 hours without further patient follow-up
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 19 | 23
milliseconds | 479.50 (42.43) | 507.80 (77.83)

3. Secondary Outcome: Controlled Oral Word Association Test
Description: The Controlled Oral Word Association Test is a measure of the ability to orally generate words to a phonemic cue within a 60-second time interval. Age and education-adjusted t-scores were used as the dependent variable. A T-score of 50 is equal to the mean, with a standard deviation of 10 points. A higher T-score is a more favorable outcome.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 19 | 23
t-scores | 49.58 (9.31) | 46.91 (8.14)

4. Secondary Outcome: Wisconsin Card Sort Test
Description: The Wisconsin Card Sorting Test is a test of rule-learning and conceptual flexibility. The participant is required to learn to sort a series of cards according to one of three principles (color, form or number) based on response feedback. The age-adjusted t-score for total number of errors was used as a dependent variable. A T-score of 50 is equal to the mean, with a standard deviation of 10 points. A higher T-score is a more favorable outcome.
Time Frame: as for outcome 2
Population: sample size for DCS group is n = 18 owing to missing data from one participant.
Measure: Mean (Standard Deviation); unit: t scores
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 18 | 23
t scores | 53.50 (12.37) | 53.70 (10.73)

5. Secondary Outcome: Trails B
Description: Trails B is a measure of cognitive flexibility. The participant alternates sequencing between numbers and letters. An age and education-adjusted t-score for time to complete the exercise was used as the dependent variable. A T-score of 50 is equal to the mean, with a standard deviation of 10 points. A higher T-score is a more favorable outcome.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 19 | 23
t-scores | 52.16 (10.99) | 48.83 (9.38)

6. Secondary Outcome: Stroop
Description: The Stroop Color Word Test is a measure of selective attention and cognitive flexibility. This measure consists of three conditions: word reading, color naming and color-word naming. The interference score (t-score) was used as the dependent variable. A T-score of 50 is equal to the mean, with a standard deviation of 10 points. Higher t-scores represent a more favorable outcome.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 19 | 23
t-score | 44.68 (7.17) | 43.30 (6.67)

7. Secondary Outcome: Implicit Memory Task
Description: Participants were presented with 32 stimulus words: 16 neutral and 16 threatening words. After a filler task (crossing out 8's on a sheet of randomized numbers) participants completed a response sheet including the stems for the 32 words presented to participants (primed words) along with stems for the 32 unprimed words. Participants were instructed to write down the first word that came to mind that completes each word stem. The priming effect was determined using the difference score between the correct number of stem completions for primed versus unprimed words. This is a value determined for each participant using the following equation: correct number of stem completions for primed word minus the correct number of stem completions for unprimed words. A larger difference score indicates a stronger implicit memory.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: correct stem completions
Arm/Group | Medication | Sugar Pill
Number analyzed (Participants) | 19 | 19
correct stem completions | 3.16 (3.24) | 2.00 (3.43)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored via a standardized side effect check list in the one hour time frame after the single dose administration and prior to neuropsychological testing. No spontaneous adverse events outside of this time frame were reported.
Arm/Group | Medication | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 3/19 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication (N=19) | Sugar Pill (N=23)
Drowsiness (General disorders) | 2 (2) | 4 (4)
Tingling sensation (General disorders) | 0 (0) | 1 (1)
Feeling lightheaded (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
DCS dosing was 1 hour prior to testing, rather than 4-8; the sample had homogenous cognitive capabilities; repeatedly administering DCS may have enhanced cognitive functioning; the measures may not have adequately tapped hippocampal-based learning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes